CLINICAL TRIAL: NCT01020721
Title: Study of Gene, Inheritance Pattern and Genotype - Phenotype Correlations in South Korean Patients With Primary Congenital Glaucoma
Brief Title: The Genetic Characteristics in South Korean Patients With Primary Congenital Glaucoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Changwon Kee, Samsung Medical Center
Other Study IDs: 2008-08-070
Record Dates: First submitted 2009-11-22; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2008-08

CONDITIONS: Primary Congenital Glaucoma
Keywords: CYP1B1 gene
MeSH Terms: conditions — Hydrophthalmos

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood
  - Genomic DNA was extracted from the peripheral leukocyte of all subjects through peripheral blood sampling
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Glaucoma: South korean patients with primary congenital glaucoma

SUMMARY:
Primary congenital glaucoma, which presents at birth or in infancy, if left untreated, may threaten vision. The incidence of congenital glaucoma varies among different geographic locations and ethnic groups.

Three genetic loci for primary congenital glaucoma (GLC3A in 2p21, GLC3B in 1p36, GLC3C in 14q24.3) were identified. CYP1B1 (cytochrome P450 1B1 ) gene, in the GLC3A locus is the main known gene and different CYP1B1 mutations has been described.

The genetic characteristics in south Korean patients with primary congenital glaucoma have not been reported yet and the genotype-phenotype correlations, the prognosis and the genetic counseling have not also been established. This study represents the first repot about the rate of CYP1B1 mutations, the genotype-phenotype correlations in south Korean patients with primary congenital glaucoma.

Patients with primary congenital glaucoma and their family will be analyzed for CYP1B1 mutations by direct sequencing of polymerase chain reaction fragments. Primary congenital glaucoma will be diagnosed according to the clinical parameters by glaucoma specialists. Patients were classified to several groups according to the pattern of mutations. Clinical parameters and genotype correlation will be compared between groups

DETAILED DESCRIPTION:
The incidence of congenital glaucoma varies among different geographic locations and ethnic group. The incidence of primary congenital glaucoma is supposed to be 0.01-0.03% in Western countries but it is reported higher in the Middle East. The inheritance pattern for congenital glaucoma is most commonly autosomal recessive. But the fact that sex distribution is unequal and the reduced penetration is seen in patients with family history implies that it's inheritance pattern is unclear. Approximately 10-40% patients have family background and the rate of penetration is known to about 10-40%.

Linkage studies have been genetic heterogeneity and have mapped three loci for primary congenital glaucoma (GLC3A in 2p21, GLC3B in 1p36, GLC3C in 14q24.3). Molecular screening of the gene or primary congenital glaucoma families liked to the 2p21 locus has determined that mutations in the cytochrome P450 1B1 (CYP1B1)are responsible for phenotype.

The genetic characteristics in south Korean patients with primary congenital glaucoma have not been not reported yet and the genotype-phenotype correlations, prognosis, genetic counseling have not established. So In this study, we evaluate the rate of CYP1B1 mutations in south Korean patients with primary congenital glaucoma and establish genotype-phenotype correlations.

Patients with primary congenital glaucoma and their family will be analyzed for CYP1B1 mutations by direct sequencing of polymerase chain reaction fragments. 100 ethnically matched normal individuals served as control subjects. Primary congenital glaucoma will be determined by examinations with slit lamp biomicroscopy, gonioscopy, measurement of intraocular pressure, corneal diameter and axial length, optic disc evaluation by glaucoma specialists. Patients were classified to several groups according to the pattern of mutations. Clinical parameters and genotype correlation will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary congenital glaucoma
* Candidate for peripheral blood sampling

Exclusion Criteria:

* Congenital glaucoma which relates with other systemic disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary congenital glaucoma who visit the glaucoma clinic in south Korea
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-03 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
clinical parameters of primary congenital glaucoma (age, onset time, symptom, intraocular pressure, corneal diameter, cup to disc ratio, axial length, treatment type) | March 2010

SECONDARY OUTCOMES:
clinical parameters of primary congenital glaucoma (age, onset time, symptom, intraocular pressure, corneal diameter, cup to disc ratio, refraction, axial length, treatment type) | september, 2010

CONTACTS AND LOCATIONS:
Overall Officials: Chang Won Kee, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Sarfarazi M, Stoilov I. Molecular genetics of primary congenital glaucoma. Eye (Lond). 2000 Jun;14 ( Pt 3B):422-8. doi: 10.1038/eye.2000.126. PMID 11026969
- [Background] Panicker SG, Mandal AK, Reddy AB, Gothwal VK, Hasnain SE. Correlations of genotype with phenotype in Indian patients with primary congenital glaucoma. Invest Ophthalmol Vis Sci. 2004 Apr;45(4):1149-56. doi: 10.1167/iovs.03-0404. PMID 15037581
- [Background] Ho CL, Walton DS. Primary congenital glaucoma: 2004 update. J Pediatr Ophthalmol Strabismus. 2004 Sep-Oct;41(5):271-88; quiz 300-1. doi: 10.3928/01913913-20040901-11. PMID 15478740
- [Background] Miller SJ. Genetic aspects of glaucoma. Trans Ophthalmol Soc U K (1962). 1966;86:425-34. No abstract available. PMID 5226587
- [Background] Gencik A. Epidemiology and genetics of primary congenital glaucoma in Slovakia. Description of a form of primary congenital glaucoma in gypsies with autosomal-recessive inheritance and complete penetrance. Dev Ophthalmol. 1989;16:76-115. PMID 2676634